CLINICAL TRIAL: NCT06687122
Title: Additional Daily Intake of Eggs for Improving Metabolic Outcomes and Choline Levels in Individuals With Obesity: Phase I Study
Brief Title: Egg Intake, Metabolic Outcomes and Choline Levels
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Guelph (Other)
Collaborators: Institut universitaire de cardiologie et de pneumologie de Québec, University Laval (Other)
Responsible Party: Principal Investigator, Clara Cho, Assistant Professor, University of Guelph
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 056099
Record Dates: First submitted 2024-11-10; First posted 2024-11-13 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Obesity and Obesity-related Medical Conditions
Keywords: Eggs; Liver health; Obesity; Metabolism; Gut microbiome
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 4 weeks of additional daily intake of 3 whole eggs (Experimental): No intervention: 4 weeks of habitual diet without daily intake of eggs (baseline) will be followed by 4 weeks of additional daily intake of 3 whole eggs then no intervention: 4 weeks of habitual diet without daily intake of eggs (washout)
  Interventions: Dietary Supplement: 3 whole eggs

INTERVENTIONS:
Dietary Supplement: 3 whole eggs — Participants will be free-living and will not be supplied with any other food except for the eggs during the intervention period with no restrictions of energy intake.

SUMMARY:
The purpose of this research is to determine the effect of additional daily egg intake on metabolic phenotypes and metabolism in the context of obesity.

DETAILED DESCRIPTION:
Choline-derived phosphatidylcholine has diverse functions including being necessary for packaging and exporting triglycerides from the liver. Choline deficiency induces fatty liver, which occurs very commonly in overweight and obesity, emphasizing the importance of choline in lipid metabolism. Studies suggest the role of gut microbiota and host genetics in influencing choline availability, which gut microbes can convert choline to trimethylamine, and hepatically oxidized by flavin monooxygenase 3 to trimethylamine-N-oxide (TMAO), a recently emerged marker of disease. We have recently shown that phosphatidylcholine (the major form of choline in food) leads to higher plasma concentrations of choline without raising TMAO compared to no choline control, which metabolic heterogeneity in TMAO response that appears to be a function of individual gut microbiota composition. However, the effect of phosphatidylcholine on parameters of liver health and function in the context of obesity has not been examined. This study will leverage a whole-food approach using eggs, which are enriched in phosphatidylcholine, as a modulator of metabolic health with a focus on interindividual variation in response.

The study objectives are: 1) determine the effect of additional daily intake of eggs on metabolic outcomes (liver density and enzymes, circulating lipids and glucose levels, body mass index and adiposity); 2) assess the effects of additional daily intake of eggs on levels of choline and downstream metabolites including TMAO; 3) determine the relation between outcome variables in response to additional daily intake of eggs and metabolic modifiers including the gut microbiota composition and genetic polymorphism. To achieve these objectives, Phase I of the larger study will be conducted, which will have multiple "hits" to form the basis of targetable outcomes. Participants will be asked to keep their habitual diet during the 4-week baseline period, followed by 4 weeks of additional daily intake of 3 whole eggs (intervention) then 4 weeks without daily intake of eggs as a washout. Participants will be free-living and will not be supplied with any other food except for the eggs during the intervention period with no restrictions of energy intake. Participants will make clinic visits every 4 weeks for 12 weeks. At their first visit (week 0), before the intervention (week 4), after the intervention (week 8) and after the washout (week 12), participants will arrive overnight-fasted and liver imaging will be performed. Fasting blood will be obtained by a phlebotomist using a standard venipuncture procedure. Anthropometric measures including waist and hip circumferences and BMI will be collected. Participants will also be asked to turn in their fecal sample in a thermos-insulated bag with ice packs. All samples will be de-identified, distributed among storage vials and stored at -80°C until further analyses.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participant of any race or ethnicity between 30-65 (inclusive) years of age
* BMI > 30 kg/m2
* Non-smoker
* Willing to consume 3 eggs per day for one dietary period of 4 weeks
* Willing to avoid eggs during the rest of the study except for eggs that are provided
* Willing to follow the study protocol including maintaining usual lifestyle during the entire study

Exclusion Criteria:

* Age < 30 or > 65 years
* BMI < 30 kg/m2
* Vegans or individuals who do not consume eggs
* Individuals who are currently pregnant or planning to become pregnant during the course of the study; or are currently breastfeeding
* Smokers, users of recreational drugs
* Individuals taking antibiotics or natural health products including prebiotics or probiotics

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-01-24 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Liver physical density by imaging technologies | Weeks 0, 4, 8 and 12
Liver morphology as assessed by imaging technologies | Weeks 0, 4, 8 and 12
Concentration of circulating liver enzymes | Weeks 0, 4, 8 and 12
Concentration of circulating lipid markers | Weeks 0, 4, 8 and 12
Concentration of circulating glucose markers | Weeks 0, 4, 8 and 12
Body mass index in kg/m^2 | Weeks 0, 4, 8 and 12
Body circumference in metrics | Weeks 0, 4, 8 and 12

SECONDARY OUTCOMES:
Choline metabolite response | Weeks 0, 4, 8 and 12
Trimethylamine-N-oxide metabolite response | Weeks 0, 4, 8 and 12
Flavin monooxygenase 3 (FMO3) 472 G>A genetic polymorphism | Week 0
Composition of fecal microbiota | Weeks 0, 4, 8 and 12

CONTACTS AND LOCATIONS:
Locations (1):
- Research Center of the Institut universitaire de cardiologie et de pneumologie de Québec - ULaval, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No
Unidentified study data can be requested for sharing within reason.

REFERENCES:
- [Background] Noga AA, Zhao Y, Vance DE. An unexpected requirement for phosphatidylethanolamine N-methyltransferase in the secretion of very low density lipoproteins. J Biol Chem. 2002 Nov 1;277(44):42358-65. doi: 10.1074/jbc.M204542200. Epub 2002 Aug 21. PMID 12193594
- [Background] Hebbard L, George J. Animal models of nonalcoholic fatty liver disease. Nat Rev Gastroenterol Hepatol. 2011 Jan;8(1):35-44. doi: 10.1038/nrgastro.2010.191. Epub 2010 Nov 30. PMID 21119613
- [Background] Zeisel SH, Da Costa KA, Franklin PD, Alexander EA, Lamont JT, Sheard NF, Beiser A. Choline, an essential nutrient for humans. FASEB J. 1991 Apr;5(7):2093-8. PMID 2010061
- [Background] Divella R, Mazzocca A, Daniele A, Sabba C, Paradiso A. Obesity, Nonalcoholic Fatty Liver Disease and Adipocytokines Network in Promotion of Cancer. Int J Biol Sci. 2019 Jan 1;15(3):610-616. doi: 10.7150/ijbs.29599. eCollection 2019. PMID 30745847
- [Background] Wang Z, Klipfell E, Bennett BJ, Koeth R, Levison BS, Dugar B, Feldstein AE, Britt EB, Fu X, Chung YM, Wu Y, Schauer P, Smith JD, Allayee H, Tang WH, DiDonato JA, Lusis AJ, Hazen SL. Gut flora metabolism of phosphatidylcholine promotes cardiovascular disease. Nature. 2011 Apr 7;472(7341):57-63. doi: 10.1038/nature09922. PMID 21475195
- [Background] Tang WH, Wang Z, Levison BS, Koeth RA, Britt EB, Fu X, Wu Y, Hazen SL. Intestinal microbial metabolism of phosphatidylcholine and cardiovascular risk. N Engl J Med. 2013 Apr 25;368(17):1575-84. doi: 10.1056/NEJMoa1109400. PMID 23614584
- [Background] Cho CE, Taesuwan S, Malysheva OV, Bender E, Tulchinsky NF, Yan J, Sutter JL, Caudill MA. Trimethylamine-N-oxide (TMAO) response to animal source foods varies among healthy young men and is influenced by their gut microbiota composition: A randomized controlled trial. Mol Nutr Food Res. 2017 Jan;61(1). doi: 10.1002/mnfr.201600324. Epub 2016 Aug 3. PMID 27377678
- [Background] Cho CE, Aardema NDJ, Bunnell ML, Larson DP, Aguilar SS, Bergeson JR, Malysheva OV, Caudill MA, Lefevre M. Effect of Choline Forms and Gut Microbiota Composition on Trimethylamine-N-Oxide Response in Healthy Men. Nutrients. 2020 Jul 25;12(8):2220. doi: 10.3390/nu12082220. PMID 32722424